CLINICAL TRIAL: NCT00253565
Title: A Phase I Dose Escalation Study of Imatinib Mesylate (Gleevec/STI571) Plus Capecitabine (Xeloda) in Advanced Solid Tumor Malignancies
Brief Title: Imatinib Mesylate and Capecitabine in Treating Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Herbert Hurwitz (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Herbert Hurwitz, Associate Professor, Duke University
Organization: Duke University (Other)
Purpose: Treatment
Other Study IDs: Pro00009521; DUMC-3992-05-8R3; ROCHE-DUMC-3992-05-8R3; NOVARTIS-DUMC-3992-05-8R3; CDR0000448905 (Other: NCI)
Record Dates: First submitted 2005-11-11; First posted 2005-11-15 (Estimated); Last update posted 2013-04-08 (Estimated); Status verified 2013-04

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — Capecitabine; Imatinib Mesylate

INTERVENTIONS:
Drug: capecitabine
Drug: imatinib mesylate

SUMMARY:
RATIONALE: Imatinib mesylate may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor. Drugs used in chemotherapy, such as capecitabine, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving imatinib mesylate together with capecitabine may kill more tumor cells.

PURPOSE: This phase I trial is studying the side effects and best dose of imatinib mesylate when given together with capecitabine in treating patients with advanced solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the maximum tolerated dose and recommended phase II dose of imatinib mesylate when administered with capecitabine in patients with advanced malignant solid tumors.

Secondary

* Determine the non-dose-limiting toxic effects of this regimen in these patients.
* Determine, preliminarily, the clinical activity of this regimen in these patients.
* Determine the pharmacokinetics and pharmacogenetics of this regimen in these patients.
* Determine, preliminarily, the effect of this regimen on wound angiogenesis in these patients.
* Correlate pharmacokinetic parameters with clinical toxicity, clinical activity, or surrogate biomarker activity of this regimen in these patients.

OUTLINE: This is a dose escalation study of imatinib mesylate.

Patients receive oral capecitabine twice daily on days 1-14 and oral imatinib mesylate once or twice daily on days 1-21. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

Cohorts of patients receive escalating doses of imatinib mesylate until the maximum tolerated dose is determined.

PROJECTED ACCRUAL: A total of 42 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed malignant solid tumors for which no standard effective therapy exists OR such therapy is refused
* Previously treated brain metastases that are currently asymptomatic allowed

PATIENT CHARACTERISTICS:

Performance status

* Karnofsky 70-100%

Life expectancy

* Not specified

Hematopoietic

* Absolute neutrophil count > 2,000/mm^3
* Platelet count > 100,000 mm^3
* Hemoglobin > 9.0 g/dL

Hepatic

* Alkaline phosphatase < 2.5 times upper limit of normal (ULN)
* SGOT and SGPT < 2.5 times ULN
* Bilirubin < 1.5 times ULN

Renal

* Creatinine clearance > 50 mL/min

Cardiovascular

* No congestive heart failure
* No symptomatic coronary artery disease
* No uncontrolled cardiac arrhythmias
* No myocardial infarction within the past 12 months
* No other clinically significant cardiac disease

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 3 months after completion of study treatment
* No prior unanticipated severe reaction to fluoropyrimidine therapy
* No known sensitivity to fluorouracil

PRIOR CONCURRENT THERAPY:

Biologic therapy

* More than 28 days since prior biologic therapy

Chemotherapy

* More than 28 days since prior chemotherapy (42 days for nitrosoureas or mitomycin C)

Endocrine therapy

* At least 90 days since prior steroids for the treatment of brain metastases
* More than 28 days since prior hormonal therapy

Radiotherapy

* At least 90 days since prior radiotherapy for the treatment of brain metastases
* More than 28 days since other prior radiotherapy
* No prior pelvic radiotherapy > 30% of the bone marrow

Surgery

* More than 28 days since prior surgery and recovered

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2003-08; Primary Completion 2006-07 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Herbert I. Hurwitz, MD, Study Chair — Duke Cancer Institute
Locations (1):
- Duke Comprehensive Cancer Center, Durham, North Carolina, United States

REFERENCES:
- [Result] Dugan E, Truax R, Meadows KL, Nixon AB, Petros WP, Favaro J, Fernando NH, Morse MA, Blobe GC, Hurwitz HI. A phase I dose-escalation study of imatinib mesylate (Gleevec/STI571) plus capecitabine (Xeloda) in advanced solid tumors. Anticancer Res. 2010 Apr;30(4):1251-6. PMID 20530436